CLINICAL TRIAL: NCT01570036
Title: Combination Immunotherapy With Herceptin and the HER2 Vaccine E75 in Low and Intermediate HER2-expressing Breast Cancer Patients to Prevent Recurrence
Brief Title: Combination Immunotherapy With Herceptin and the HER2 Vaccine NeuVax
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: George E. Peoples (Industry)
Collaborators: Genentech, Inc. (Industry); Sellas Life Sciences Group (Industry)
Responsible Party: Sponsor-Investigator, George E. Peoples, President and CEO, Cancer Insight, LLC, Cancer Insight, LLC
Organization: Cancer Insight, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 368255; 1137008 / 20130058 (Other: Western Institutional Review Board)
Record Dates: First submitted 2012-03-25; First posted 2012-04-04 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; HER2 peptide (369-377); Receptor Protein-Tyrosine Kinases; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Herceptin + NeuVax vaccine (Experimental): Patients randomized to this arm will receive Herceptin every 3 weeks as monotherapy for 1 year; the first Herceptin infusion will be given no sooner than 3 weeks and no later than 12 weeks after completion of standard of care chemotherapy/radiotherapy. Herceptin will be dosed at the recommended initial loading dose of 8 mg/kg and at recommended maintenance doses of 6 mg/kg q3wk. Patients will receive vaccinations of NeuVax vaccine administered intradermally every 3 weeks for 6 total vaccinations, 30-120 minutes after completion of Herceptin infusion. The NeuVax vaccine series will begin immediately after completion of the third Herceptin infusion, but may be delayed to the fourth or fifth Herceptin infusion with prior approval from the PI. Patients will be blinded regarding assigned arm. After completion of primary vaccine series, patients will receive 4 NeuVax vaccine booster inoculations to be administered every 6 months x 4 for total treatment duration of 30 months.
  Interventions: Drug: Herceptin; Drug: NeuVax vaccine; Drug: GM-CSF
- Herceptin + GM-CSF only (Active Comparator): Patients randomized to this arm will receive Herceptin every 3 weeks as monotherapy for 1 year. The first Herceptin infusion will be given no sooner than 3 weeks and no later than 12 weeks after completion of standard of care chemotherapy/radiotherapy. Herceptin will be dosed at the recommended initial loading dose of 8 mg/kg and at recommended maintenance doses of 6 mg/kg q3wk. Patients will receive inoculations of GM-CSF only (250mcg) administered intradermally every 3 weeks for 6 total inoculations, 30-120 minutes after completion of Herceptin infusion. The GM-CSF only inoculation series will begin immediately after completion of the third Herceptin infusion. Patients will be blinded as to whether they are receiving NeuVax vaccine or GM-CSF only. After completion of six-inoculation primary vaccine series, patients will then receive a total of four GM-CSF only booster inoculations to be administered at 12, 18, 24, and 30 months from the date of the first Herceptin infusion.
  Interventions: Drug: Herceptin; Drug: GM-CSF

INTERVENTIONS:
Drug: Herceptin — Herceptin will be administered to patients every three weeks as monotherapy for one year, to be given upon completion of standard of care chemotherapy/radiotherapy. The first Herceptin infusion will be given no sooner than three weeks and no later than 12 weeks after completion of chemotherapy/radiotherapy. Herceptin will be dosed at the recommended initial loading dose of 8 mg/kg and at recommended maintenance doses of 6 mg/kg q3wk.
  Other Names: Trastuzumab
Drug: NeuVax vaccine — At the time of vaccine administration, a frozen solution of E75 acetate (1.5mg/ml) is thawed and 1000mcg E75 peptide mixed thoroughly with 250mcg GM-CSF. This constitutes the NeuVax vaccine. For patients randomized to the Herceptin + NeuVax vaccine arm, they will commence Herceptin monotherapy and then will begin the NeuVax vaccine series immediately after completion of the third Herceptin infusion. The vaccine series consists of NeuVax vaccine administered intradermally every three weeks for six total vaccinations, 30-120 minutes after completion of Herceptin infusion.
  Other Names: E75 peptide (KIFGSLAFL, HER2/neu, 369-377); GM-CSF (sargramostim)
  Arms: Herceptin + NeuVax vaccine
Drug: GM-CSF — For patients randomized to the Herceptin + GM-CSF only arm, they will commence Herceptin monotherapy and then will begin the GM-CSF inoculation series immediately after completion of the third Herceptin infusion. The GM-CSF inoculation series consists of 250mcg GM-CSF administered intradermally every three weeks for six total vaccinations, 30-120 minutes after completion of Herceptin infusion.
  Other Names: Sargramostim

SUMMARY:
The study will be a multi-center, prospective, randomized, single-blinded, placebo-controlled Phase II trial of Herceptin + NeuVax(TM) vaccine (E75 peptide/granulocyte macrophage-colony stimulating factor) (GM-CSF) versus Herceptin + GM-CSF alone. The target study population is node-positive (NP) (or node-negative [NN] if negative for both ER and PR) breast cancer patients with HER2 1+ and 2+ expressing tumors who are disease-free after standard of care therapy. Disease-free subjects after standard of care multi-modality therapy will be screened and HLA-typed. E75 is a CD8-eliciting peptide vaccine that was restricted to HLA-A2+ or HLA-A3+ patients (approximately two-thirds of the US population), and has been extended to HLA-A24+ and HLA-A26+ as well.

DETAILED DESCRIPTION:
In this study, the investigators intend to assess the ability of the combination of Herceptin and NeuVax vaccine (HER2 protein E75 peptide administered with the immunoadjuvant GM-CSF) given in the adjuvant setting to prevent recurrences in NP (or NN if negative for both estrogen (ER) and progesterone (PR) receptors) breast cancer patients with tumors that express low (1+) or intermediate (2+) levels of HER2. Enrolled patients will be randomized to receive Herceptin and NeuVax vaccine or Herceptin with GM-CSF alone (no NeuVax vaccine). The safety of the combination therapy will be documented, specifically to ensure that no additive cardiac toxicity results from combination HER2-directed therapy. Efficacy will be documented by comparing the DFS and immunological responses between treatment groups.

The primary efficacy endpoint is to compare DFS at 24 months between treatment groups. The primary safety issue is to prove there is no additive cardiac toxicity with combination HER2-directed therapy. A secondary endpoint of the trial is to compare DFS at 36 months. Immunologic responses to the vaccine will also be documented and correlated to clinical benefit.

The study will be a multi-center, prospective, randomized, single-blinded, placebo-controlled Phase II trial of Herceptin + NeuVax vaccine versus Herceptin + GM-CSF alone. The target study population is NP (or NN if negative for both ER and PR) breast cancer patients with HER2 1+ and 2+ expressing tumors who are disease-free after standard of care therapy. Disease-free subjects after standard of care multi-modality therapy will be screened and HLA-typed. E75 is a CD8-eliciting peptide vaccine that is restricted to HLA-A2+ or HLA-A3+ patients (approximately two-thirds of the US population), and has been extended to HLA-A24+ and HLA-A26+ as well.

HLA-A2+/A3+/A24+/or A26+ patients who meet all other eligibility criteria will be randomized to receive Herceptin + NeuVax vaccine or Herceptin + GM-CSF alone. For both groups, Herceptin will be given every three weeks as monotherapy for one year, to be given upon completion of standard of care chemotherapy/radiotherapy. The first Herceptin infusion must be given no sooner than three weeks and no later than 12 weeks after completion of chemotherapy/radiotherapy. Herceptin will be dosed at the recommended initial loading dose of 8 mg/kg and at recommended maintenance doses of 6 mg/kg q3wk. Herceptin will be administered as described in Section 4.3. Patients randomized to the NeuVax vaccine arm will receive vaccinations of E75 peptide (1000 mcg) and GM-CSF (250 mcg) administered intradermally every three weeks for six total vaccinations, 30-120 minutes after completion of Herceptin infusion. The NeuVax vaccine series will begin immediately after completion of the third Herceptin infusion. In extenuating circumstances, the first vaccination may be delayed to the fourth or fifth Herceptin infusion with prior approval from the Principal Investigator. Those patients randomized to the GM-CSF alone arm will receive vaccinations of GM-CSF (250 mcg) administered in an identical manner to those receiving NeuVax vaccine. Patients will be blinded as to whether they are receiving NeuVax vaccine or GM-CSF alone.

Upon completion of the vaccination series, booster inoculations (same dose and route) will be administered every six months x4 for total combination (Herceptin and vaccine) treatment duration of 30 months. The first booster inoculation will occur with the final Herceptin infusion, with subsequent boosters timed every six months from the first booster. Booster inoculations will occur for patients randomized to receive E75/GM-CSF as well as patients randomized to receive GM-CSF alone, and will consist of the same treatment drugs and dosing (i.e. E75/GM-CSF patients will be boosted with E75/GM-CSF while GM-CSF alone patients will be boosted with GM-CSF alone). Patient blinding will be maintained throughout the study.

Subjects will be followed for safety issues, immunologic response and clinical recurrence. Patients will be monitored 48-72 hours after each inoculation for reaction to the inoculation as well as documentation of any adverse effects experienced. Immunologic response will be documented with both in vitro phenotypic and functional assays as well as in vivo delayed type hypersensitivity (DTH) reactions. All patients will be followed for a total of 36 months to document disease-free status.

The investigators plan to enroll 300 patients (150 in each treatment arm) at a planned accrual rate of 12 patients per month (approximately one per study site per month). With accrual beginning in April, 2013, enrollment of the last patient would be expected in August 2017 followed by a three-year follow-up period. The duration of the trial is expected to be seven years.

ELIGIBILITY:
Patients will be included in the study based on the following criteria:

* Women 18 years or older
* Node-positive breast cancer (AJCC N1, N2, or N3)
* Node-negative breast cancer if negative for both estrogen (ER) and progesterone (PR) receptors and have received chemotherapy as standard of care
* Clinically cancer-free (no evidence of disease) after standard of care therapy (surgery, chemotherapy, radiation therapy as directed by NCCN guidelines). Hormonal therapy will continue per standard of care. Neoadjuvant chemotherapy is allowed.
* Recovery from any toxicity(ies) associated with prior adjuvant therapy.
* HER2 expression of 1+ or 2+ by IHC. FISH or Dual-ISH testing must be performed on IHC 2+ tumors and shown to be non-amplified by FISH (≤2.0) or by Dual-ISH (≤2.0).
* HLA-A2, A3, A24, or A26 positive
* LVEF >50%, or an LVEF within the normal limits of the institution's specific testing (MUGA or Echo)
* ECOG 0,1
* Signed informed consent
* Adequate birth control (abstinence, hysterectomy, bilateral oophorectomy, bilateral tubal ligation, oral contraception, IUD, or use of condoms or diaphragms)
* Must start study treatment (receive first Herceptin infusion) 15between 3-12 weeks from completion of standard of care therapy.

4.1.3 Exclusion Criteria

Patients will be excluded from the study based on the following criteria:

* Node-negative breast cancer (AJCC N0 or N0(i+)) unless negative for both estrogen (ER) and progesterone (PR) receptors and has received chemotherapy as standard of care
* Clinical or radiographic evidence of distant or residual breast cancer
* HER2 negative (IHC 0) or HER2 3+ or FISHDual-ISH amplified (FISH >2.0); Dual-ISH >2.0
* HLA-A2, A3, A24, A26 negative
* History of prior Herceptin therapy
* NYHA stage 3 or 4 cardiac disease
* LVEF <50%, or less than the normal limits of the institution's specific testing (MUGA or Echo)
* Immune deficiency disease or HIV, HBV, HCV
* Receiving immunosuppressive therapy including chemotherapy, chronic steroids, methotrexate, or other known immunosuppressive agents
* ECOG ≥2
* Tbili >1.8, creatinine>2, hemoglobin<10, platelets<50,000, WBC<2,000
* Pregnancy (assessed by urine HCG)
* Breast feeding
* Any active autoimmune disease requiring treatment, with the exception of vitiligo
* Active pulmonary disease requiring medication to include multiple inhalers
* Involved in other experimental protocols (except with permission of the other study PI)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2013-05-21 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: COL (ret.) George E. Peoples, MD, FACS, Principal Investigator — Cancer Insight, LLC; COL (ret.) George E. Peoples, MD, FACS, Study Director — Cancer Insight, LLC
Locations (29):
- United States (29):
  - Samuel Oschin Comprehensive Cancer Institute - Cedars Sinai Medical Center, Beverly Hills, California
  - Sarcoma Oncology Research Center, LLC, Santa Monica, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Katzen Cancer Research Center, George Washington University, Washington D.C., District of Columbia
  - University of Miami, Deerfield Beach, Florida
  - University of Miami, Kendall, Florida
  - University of Miami, Miami, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - University of Miami, Plantation, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Inc, Tampa, Florida
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Medstar Health - Union Memorial Hospital, Baltimore, Maryland
  - Medstar Health - Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - MedStar Health - Good Samaritan Hospital, Baltimore, Maryland
  - The Valley Hospital, Paramus, New Jersey
  - Tisch Cancer Institute/Icahn School of Medicine at Mount Sinai, New York, New York
  - North Shore Hematology Oncology Associates, The Bronx, New York
  - Legacy Health, Legacy Good Samaritan Medical Center, Portland, Oregon
  - Thomas Jefferson University - Kimmel Cancer Center, Philadelphia, Pennsylvania
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Texas Oncology (Cancer Care Centers of South Texas), San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Providence Regional Medical Center, Everett, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Columbia St. Mary's, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Clifton GT, Hale D, Vreeland TJ, Hickerson AT, Litton JK, Alatrash G, Murthy RK, Qiao N, Philips AV, Lukas JJ, Holmes JP, Peoples GE, Mittendorf EA. Results of a Randomized Phase IIb Trial of Nelipepimut-S + Trastuzumab versus Trastuzumab to Prevent Recurrences in Patients with High-Risk HER2 Low-Expressing Breast Cancer. Clin Cancer Res. 2020 Jun 1;26(11):2515-2523. doi: 10.1158/1078-0432.CCR-19-2741. Epub 2020 Feb 18. PMID 32071118

RESULTS

PARTICIPANT FLOW:
Groups:
- Herceptin + NeuVax Vaccine: Patients randomized to this arm will receive Herceptin every 3 weeks as monotherapy for 1 year; the first Herceptin infusion will be given no sooner than 3 weeks and no later than 12 weeks after completion of standard of care chemotherapy/radiotherapy. Herceptin will be dosed at the recommended initial loading dose of 8 mg/kg and at recommended maintenance doses of 6 mg/kg q3wk. Patients will receive vaccinations of NeuVax vaccine administered intradermally every 3 weeks for 6 total vaccinations, 30-120 minutes after completion of Herceptin infusion. The NeuVax vaccine series will begin immediately after completion of the third Herceptin infusion, but may be delayed to the fourth or fifth Herceptin infusion with prior approval from the PI. After completion of primary vaccine series, patients will receive NeuVax vaccine booster inoculations to be administered every 6 months x 4 for total treatment duration of 30 months.
- Herceptin + GM-CSF Only: Patients randomized to this arm will receive Herceptin every 3 weeks as monotherapy for 1 year. The first Herceptin infusion will be given no sooner than 3 weeks and no later than 12 weeks after completion of standard of care chemotherapy/radiotherapy. Herceptin will be dosed at the recommended initial loading dose of 8 mg/kg and at recommended maintenance doses of 6 mg/kg q3wk. Patients will receive inoculations of GM-CSF only (250mcg) administered intradermally every 3 weeks for 6 total inoculations, 30-120 minutes after completion of Herceptin infusion. The GM-CSF only inoculation series will begin immediately after completion of the third Herceptin infusion. After completion of six-inoculation primary vaccine series, patients will then receive a total of four GM-CSF only booster inoculations to be administered at 12, 18, 24, and 30 months from the date of the first Herceptin infusion.
Period: Overall Study
Arm/Group | Herceptin + NeuVax Vaccine | Herceptin + GM-CSF Only
Started | 136 | 139
Primary Vaccine Series Completed | 121 | 132
Booster Series Completed | 40 | 30
Completed | 18 | 17
Not Completed | 118 | 122

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Herceptin + NeuVax Vaccine | Herceptin + GM-CSF Only | Total
Number analyzed (Participants) | 136 | 139 | 275
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52.2 [43.7 to 60.8] | 50.5 [42 to 59] | 51.6 [43.9 to 61.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 139 | 275
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 109 | 97 | 206
  Asian | 2 | 9 | 11
  Black | 13 | 20 | 33
  Hispanic | 10 | 9 | 19
  Unknown | 2 | 4 | 6
Nottingham modified, Scarff-Bloom-Richardson Grade [Count of Participants; unit: Participants] — Pathological grading system based on tumor tubule formation, number of mitotic figures in most active areas and nuclear pleomorphism. Each of these factors is given points 1-3 for a total of 3-9 points. The overall scores are broken down as 3 - 5 points (well differentiated (grade I)), 6 - 7 points (moderately differentiated (grade II)), and 8 - 9 points (poorly differentiated (grade III)).
  Participants
    Grade 1 | 8 | 14 | 22
    Grade 2 | 57 | 56 | 113
    Grade 3 | 69 | 69 | 138
Hormone receptor status [Count of Participants; unit: Participants]
  ER Positive | 81 | 95 | 176
  PR Positive | 77 | 83 | 160
  Triple Negative | 53 | 44 | 97
HER2 Immunohistochemistry (IHC) [Count of Participants; unit: Participants] — IHC 1+ is incomplete membrane staining that is faint/barely perceptible and within >10% of the invasive tumor cells. IHC 2+ is a weak to moderate complete membrane staining is observed in >10% of tumor cells OR strong complete membrane staining in </= 10% of tumor cells.
  Participants
    IHC 1+ | 89 | 89 | 178
    IHC 2+ | 47 | 50 | 97
Breast surgery [Count of Participants; unit: Participants]
  Breast Conservation Therapy | 39 | 34 | 73
  Mastectomy | 97 | 104 | 201
  None | 0 | 1 | 1
Chemotherapy [Count of Participants; unit: Participants]
  Neoadjuvant | 72 | 76 | 148
  Adjuvant | 59 | 57 | 116
  None | 5 | 6 | 11
Radiation with Breast Conservation Therapy [Count of Participants; unit: Participants] — Population: Only evaluable for patients that underwent breast conservation therapy.
  Participants
    Adjuvant: number analyzed (Participants) | 39 | 34 | 73
    Adjuvant | 39 | 34 | 73
    None: number analyzed (Participants) | 39 | 34 | 73
    None | 0 | 0 | 0
Radiation with Mastectomy [Count of Participants; unit: Participants] — Population: Only evaluable for patients that underwent mastectomy.
  Participants
    Adjuvant: number analyzed (Participants) | 97 | 104 | 201
    Adjuvant | 76 | 89 | 165
    Neoadjuvant: number analyzed (Participants) | 97 | 104 | 201
    Neoadjuvant | 2 | 0 | 2
    None: number analyzed (Participants) | 97 | 104 | 201
    None | 19 | 15 | 34
Axillary Surgery [Count of Participants; unit: Participants]
  Axillary Dissection | 81 | 88 | 169
  Sentinel Lymph Node Biopsy | 55 | 48 | 103
  None | 0 | 3 | 3
AJCC, 7th Edition, Clinical Stage (for patients receiving neoadjuvant chemotherapy) [Count of Participants; unit: Participants] — Stage 0 is not cancer, abnormal cells are present but not spread Stage I-III Cancer is present. The higher number, the larger tumor & more spread to nearby tissues Stage IV Cancer has distant body part spread(AJCC, 7th Ed) Clinical staging occurs prior to neoadjuvant chemo Only neoadjuvant chemotherapy patients included
  *1 patient with path. stage IIB after completion of chemo was enrolled & vaccinated. It was discovered the patient had metastatic disease prior to initiation chemotherapy & enrolled in protocol violation. The patient was in eligible & excluded from efficacy analyses. Population: Only neoadjuvant chemotherapy patients included into this patient count.
  Participants
    Unknown: number analyzed (Participants) | 72 | 76 | 148
    Unknown | 1 | 2 | 3
    0: number analyzed (Participants) | 72 | 76 | 148
    0 | 0 | 1 | 1
    I: number analyzed (Participants) | 72 | 76 | 148
    I | 4 | 3 | 7
    IIA: number analyzed (Participants) | 72 | 76 | 148
    IIA | 16 | 13 | 29
    IIB: number analyzed (Participants) | 72 | 76 | 148
    IIB | 19 | 18 | 37
    IIIA: number analyzed (Participants) | 72 | 76 | 148
    IIIA | 14 | 25 | 39
    IIIB: number analyzed (Participants) | 72 | 76 | 148
    IIIB | 7 | 2 | 9
    IIIC: number analyzed (Participants) | 72 | 76 | 148
    IIIC | 10 | 13 | 23
    IV*: number analyzed (Participants) | 72 | 76 | 148
    IV* | 1 | 0 | 1
AJCC, 7th Edition, Pathologic Stage (for patients receiving neoadjuvant chemotherapy) [Count of Participants; unit: Participants] — Stage 0 is not cancer, abnormal cells are present but not spread Stage I-III Cancer is present. The higher number, the larger tumor & more spread to nearby tissues Stage IV Cancer has distant body part spread
  The American Joint Committee on Cancer, 7th Edition Staging was used for this analysis (https://cancerstaging.org/references-tools/quickreferences/Documents/BreastMedium.pdf).
  Pathologic staging occurs after patients have undergone surgical therapy.
  Only neoadjuvant chemotherapy patients included into this patient count. Population: Only neoadjuvant chemotherapy patients included into this patient count.
  Participants
    Unknown: number analyzed (Participants) | 72 | 76 | 148
    Unknown | 1 | 0 | 1
    0: number analyzed (Participants) | 72 | 76 | 148
    0 | 5 | 4 | 9
    I: number analyzed (Participants) | 72 | 76 | 148
    I | 11 | 9 | 20
    IIA: number analyzed (Participants) | 72 | 76 | 148
    IIA | 16 | 15 | 31
    IIB: number analyzed (Participants) | 72 | 76 | 148
    IIB | 12 | 11 | 23
    IIIA: number analyzed (Participants) | 72 | 76 | 148
    IIIA | 11 | 20 | 31
    IIIB: number analyzed (Participants) | 72 | 76 | 148
    IIIB | 4 | 3 | 7
    IIIC: number analyzed (Participants) | 72 | 76 | 148
    IIIC | 12 | 14 | 26
AJCC, 7th Edition, Pathologic Stage [Count of Participants; unit: Participants] — Stage 0 is not cancer, abnormal cells are present but not spread Stage I-III Cancer is present. The higher number, the larger tumor & more spread to nearby tissues Stage IV Cancer has distant body part spread
  The American Joint Committee on Cancer, 7th Edition Staging was used for this analysis (https://cancerstaging.org/references-tools/quickreferences/Documents/BreastMedium.pdf).
  Pathologic staging is performed after the patients have undergone surgical therapy; these patient did not receive neoadjuvant chemotherapy. Population: The analysis only includes patients that did not receive neoadjuvant chemotherapy (thus, adjuvant and none).
  Participants
    I: number analyzed (Participants) | 64 | 63 | 127
    I | 10 | 9 | 19
    IIA: number analyzed (Participants) | 64 | 63 | 127
    IIA | 11 | 12 | 23
    IIB: number analyzed (Participants) | 64 | 63 | 127
    IIB | 14 | 14 | 28
    IIIA: number analyzed (Participants) | 64 | 63 | 127
    IIIA | 21 | 18 | 39
    IIIB: number analyzed (Participants) | 64 | 63 | 127
    IIIB | 0 | 0 | 0
    IIIC: number analyzed (Participants) | 64 | 63 | 127
    IIIC | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: Disease-free survival (DFS) for all patients regardless of randomization will be determined by patients' own physicians at the individual study sites during routine follow-up screening. This will occur every three months for the first 24 months after completion of primary therapies and every six months thereafter with clinical exam, and laboratory and radiographic surveillance. The primary objective of the study is disease-free survival (DFS) at 24 months.
Time Frame: Disease-free survival at 24 months
Measure: Number; unit: Percentage of participants who survived
Arm/Group | Herceptin + NeuVax Vaccine | Herceptin + GM-CSF Only
Number analyzed (Participants) | 136 | 139
Percentage of participants who survived | 89.8 | 83.8
Statistical Analysis 1: Comparison: Herceptin + NeuVax Vaccine vs Herceptin + GM-CSF Only; Test type: Other — Kaplan-Meier Survival Analysis; p = 0.18, Kaplan-Meier Survival Analysis; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [.31 to 1.25]

2. Primary Outcome: Disease-free Survival (DFS)
Description: Disease-free survival (DFS) for all patients regardless of randomization will be determined by patients' own physicians at the individual study sites during routine follow-up screening. This will occur at months 30 and 36 after completion of primary therapies with clinical exam, and laboratory and radiographic surveillance. The secondary objective of the study is disease-free survival (DFS) at 36 months.
Time Frame: Disease-free survival up to 36 months
Measure: Number; unit: Percent Survival
Arm/Group | Herceptin + NeuVax Vaccine | Herceptin + GM-CSF Only
Number analyzed (Participants) | 136 | 139
Percent Survival | 86.7 | 80.8

3. Secondary Outcome: Percent Ejection Fraction - A Measure of Cardiac Toxicity
Description: Each patient, regardless of randomization, will undergo cardiac assessment (ejection fraction) of Multiple Gated Acquisition scan (MUGA) preferred, echocardiogram (ECHO) allowed, consistency required) at baseline, 3 months, 6 months, 12 months, and 24 months. Cardiac assessment will continue every six months if a patient experiences a greater than 10% reduction from baseline for the duration of the trial or until resolution.
Time Frame: 24 months
Population: The analysis was performed on those patients with data at each specified time point.
Measure: Mean (Standard Error); unit: Percent Ejection Fraction
Arm/Group | Herceptin + NeuVax Vaccine | Herceptin + GM-CSF Only
Number analyzed (Participants) | 136 | 137
Percent Ejection Fraction
  Baseline | 60.82 (.61) | 61.47 (.47)
  3 Months: number analyzed (Participants) | 126 | 121
  3 Months | 59.49 (.54) | 59.56 (.54)
  6 Months: number analyzed (Participants) | 116 | 112
  6 Months | 59.92 (.88) | 60.07 (.57)
  12 Months: number analyzed (Participants) | 96 | 87
  12 Months | 59.39 (.56) | 59.7 (.57)
  24 Months: number analyzed (Participants) | 54 | 43
  24 Months | 61.05 (.79) | 61.09 (.78)
Statistical Analysis 1: Comparison: Herceptin + NeuVax Vaccine vs Herceptin + GM-CSF Only; Test type: Other; p = 0.02, ANOVA — Comparison of the mean LVEF from baseline to 3 months, 6 months, and 12 months; this time period includes the therapy period of trastuzumab
Statistical Analysis 2: Comparison: Herceptin + NeuVax Vaccine vs Herceptin + GM-CSF Only; Test type: Other; p = 0.58, ANOVA — The mean LVEF compared at baseline to 3 months, 6 months, 12 months and 24 months; this time period includes the duration of trastuzumab therapy and 1 year after completion of trastuzumab therapy
Statistical Analysis 3: Comparison: Herceptin + NeuVax Vaccine vs Herceptin + GM-CSF Only; Test type: Other; p = 0.65, Regression, Linear — Evaluating LVEF at all time points with a linear mixed regression model, this analysis compared cardiac ejection fraction over time
Statistical Analysis 4: Comparison: Herceptin + NeuVax Vaccine vs Herceptin + GM-CSF Only; Test type: Other; p = 0.91, Regression, Linear — This analysis evaluated LVEF at all time points with a linear mixed regression model between randomization arms
Statistical Analysis 5: Comparison: Herceptin + NeuVax Vaccine vs Herceptin + GM-CSF Only; Test type: Other; p = 0.81, Regression, Linear — This analysis evaluated LVEF at all time points with a linear mixed regression model between the arms over time

4. Secondary Outcome: Local and Systemic Toxicities
Description: Standard local and systemic toxicities will be collected and graded per the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03 toxicity scale. For both the regular and booster inoculations, patients will be monitored closely for one hour after inoculation with questioning, serial exams and vital signs every 15 minutes to observe for a hypersensitivity reaction. Patients will also return to the clinic 48-72 hours after each inoculation for questioning regarding systemic toxicity and to examine and measure the local reaction at the inoculation sites. Reported are the maximum related and graded adverse events per patient.
Time Frame: Duration of vaccine or inoculation series and booster series, an average of 30 months.
Population: The safety analysis was performed only on patients that received NeuVax or Control.
Measure: Number; unit: Percent Experiencing
Arm/Group | Herceptin + NeuVax Vaccine | Herceptin + GM-CSF Only
Number analyzed (Participants) | 129 | 132
Percent Experiencing
  Local Grade 1 | 82.3 | 55.7
  Local Grade 2 | 15.0 | 33.0
  Local Grade 3 | 2.7 | 11.3
  Systemic Grade 1 | 79.6 | 58.5
  Systemic Grade 2 | 20.4 | 30.2
  Systemic Grade 3 | 0 | 11.3
Statistical Analysis 1: Comparison: Herceptin + NeuVax Vaccine vs Herceptin + GM-CSF Only; The safety group consisted of any patients who received NPS with GM-CSF or placebo with GM-CSF inoculations; Test type: Other; p = 0.149, Chi-squared; Comparison of the maximum related local toxicity experienced per patient and compared between treatment arms
Statistical Analysis 2: Comparison: Herceptin + NeuVax Vaccine vs Herceptin + GM-CSF Only; Test type: Other; p = 0.901, Chi-squared; Comparison of the maximum related systemic toxicity experienced per patient and compared between treatment arms

ADVERSE EVENTS:
Time Frame: The duration of the trial, up to 36 months.
Arm/Group | Herceptin + NeuVax Vaccine | Herceptin + GM-CSF Only
All-Cause Mortality (participants affected / at risk) | 1/136 | 0/139
Serious Adverse Events (participants affected / at risk) | 14/136 | 12/139
Other Adverse Events (participants affected / at risk) | 136 | 139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Herceptin + NeuVax Vaccine (N=136) | Herceptin + GM-CSF Only (N=139)
Skin Infection (Infections and infestations) | 1 (1) | 1 (1) — Local
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Systemic
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Systemic
Heart failure (Cardiac disorders) | 1 (1) | 1 (2) — Systemic
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Systemic
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Systemic
Esophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) — Systemic
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Systemic
Fever (General disorders) | 1 (2) | 0 (0) — Systemic
Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) — Systemic
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) — Systemic
Breast infection (Infections and infestations) | 1 (1) | 1 (1) — Systemic
Device related infection (Infections and infestations) | 0 (0) | 1 (1) — Systemic
Skin Infection (Infections and infestations) | 1 (2) | 0 (0) — Systemic
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) — Systemic
Wound infection (Infections and infestations) | 1 (1) | 0 (0) — Systemic
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Systemic
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Systemic
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Systemic
Creatinine increased (Investigations) | 0 (0) | 1 (1) — Systemic
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Systemic
Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) — Systemic
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1) — Systemic
Seizure (Nervous system disorders) | 0 (0) | 1 (1) — Systemic
Syncope (Nervous system disorders) | 1 (1) | 0 (0) — Systemic
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) — Systemic
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Systemic
Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Systemic
Thromboembolic event (Vascular disorders) | 2 (2) | 2 (2) — Systemic
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Herceptin + NeuVax Vaccine | Herceptin + GM-CSF Only
Injection site reaction (General disorders) | 109/136 (846) | 102/139 (698) — Local
Fatigue (General disorders) | 2/136 (2) | 1/139 (1) — Local
Pain (General disorders) | 49/136 (140) | 32/139 (83) — Local
Other, specify (General disorders) | 1/136 (1) | 0/139 (0) — Local
Malaise (General disorders) | 0/136 (0) | 1/139 (1) — Local
Chills (General disorders) | 1/136 (1) | 0/139 (0) — Local
Flu like symptoms (General disorders) | 0/136 (0) | 1/139 (1) — Local
Edema limbs (General disorders) | 1/136 (4) | 2/139 (3) — Local
Infusion related reaction (General disorders) | 1/136 (1) | 0/139 (0) — Local
Localized edema (General disorders) | 1/136 (1) | 1/139 (1) — Local
Facial pain (General disorders) | 0/136 (0) | 1/139 (1) — Local
Pruritus (Skin and subcutaneous tissue disorders) | 95/136 (429) | 89/139 (371) — Local
Skin induration (Skin and subcutaneous tissue disorders) | 81/136 (337) | 67/139 (244) — Local
Other, specify (Skin and subcutaneous tissue disorders) | 9/136 (13) | 10/139 (21) — Local
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1/136 (1) | 3/139 (11) — Local
Rash acneiform (Skin and subcutaneous tissue disorders) | 0/136 (0) | 1/139 (4) — Local
Nail loss (Skin and subcutaneous tissue disorders) | 0/136 (0) | 1/139 (1) — Local
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 2/136 (2) | 0/139 (0) — Local
Arthralgia (Musculoskeletal and connective tissue disorders) | 2/136 (2) | 3/139 (3) — Local
Myalgia (Musculoskeletal and connective tissue disorders) | 3/136 (5) | 8/139 (12) — Local
Other, specify (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 1/139 (1) — Local
Back pain (Musculoskeletal and connective tissue disorders) | 2/136 (7) | 2/139 (10) — Local
Bone pain (Musculoskeletal and connective tissue disorders) | 1/136 (1) | 2/139 (2) — Local
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4/136 (4) | 6/139 (11) — Local
Neck pain (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 1/139 (1) — Local
Headache (Nervous system disorders) | 5/136 (5) | 4/139 (12) — Local
Neuropathy (Nervous system disorders) | 1/136 (1) | 1/139 (1) — Local
Peripheral sensory neuropathy (Nervous system disorders) | 1/136 (1) | 2/139 (2) — Local
Dysgeusia (Nervous system disorders) | 1/136 (1) | 2/139 (2) — Local
Paresthesia (Nervous system disorders) | 1/136 (1) | 0/139 (0) — Local
Nausea (Gastrointestinal disorders) | 1/136 (1) | 2/139 (2) — Local
Other, specify (Gastrointestinal disorders) | 1/136 (1) | 2/139 (2) — Local
Diarrhea (Gastrointestinal disorders) | 0/136 (0) | 2/139 (2) — Local
Abdominal pain (Gastrointestinal disorders) | 0/136 (0) | 2/139 (2) — Local
Anal hemorrhage (Gastrointestinal disorders) | 1/136 (2) | 0/139 (0) — Local
Toothache (Gastrointestinal disorders) | 1/136 (1) | 0/139 (0) — Local
Dental abscess (Gastrointestinal disorders) | 0/136 (0) | 1/139 (1) — Local
Chelitis (Gastrointestinal disorders) | 1/136 (1) | 0/139 (0) — Local
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0/136 (0) | 2/139 (2) — Local
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/136 (1) | 0/139 (0) — Local
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2/136 (2) | 3/139 (5) — Local
Cough (Respiratory, thoracic and mediastinal disorders) | 0/136 (0) | 1/139 (1) — Local
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2/136 (2) | 2/139 (2) — Local
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/136 (0) | 1/139 (1) — Local
Breast pain (Respiratory, thoracic and mediastinal disorders) | 0/136 (0) | 1/139 (1) — Local
Upper respiratory infection (Infections and infestations) | 1/136 (2) | 1/139 (1) — Local
Sinusitis (Infections and infestations) | 1/136 (1) | 1/139 (1) — Local
Skin infection (Infections and infestations) | 3/136 (3) | 1/139 (1) — Local
Breast infection (Infections and infestations) | 1/136 (1) | 1/139 (1) — Local
Lip infection (Infections and infestations) | 0/136 (0) | 1/139 (2) — Local
Otitis media (Infections and infestations) | 1/136 (1) | 0/139 (0) — Local
Wound infection (Infections and infestations) | 1/136 (1) | 0/139 (0) — Local
Pharyngitis (Infections and infestations) | 0/136 (0) | 1/139 (1) — Local
Device related infection (Infections and infestations) | 0/136 (0) | 1/139 (1) — Local
Eye infection (Infections and infestations) | 1/136 (1) | 0/139 (0) — Local
Hot flashes (Vascular disorders) | 2/136 (2) | 1/139 (1) — Local
Lymphedema (Vascular disorders) | 0/136 (0) | 1/139 (1) — Local
Hematoma (Vascular disorders) | 1/136 (1) | 0/139 (0) — Local
White blood cell decreased (Investigations) | 0/136 (0) | 1/139 (1) — Local
Other, specify (Injury, poisoning and procedural complications) | 1/136 (1) | 1/139 (1) — Local
Bruising (Injury, poisoning and procedural complications) | 10/136 (12) | 10/139 (14) — Local
Fracture (Injury, poisoning and procedural complications) | 2/136 (2) | 0/139 (0) — Local
Seroma (Injury, poisoning and procedural complications) | 1/136 (1) | 0/139 (0) — Local
Burn (Injury, poisoning and procedural complications) | 1/136 (1) | 0/139 (0) — Local
Anxiety (Psychiatric disorders) | 0/136 (0) | 1/139 (1) — Local
Other, specify (Eye disorders) | 0/136 (0) | 1/139 (1) — Local
Watering eyes (Eye disorders) | 0/136 (0) | 2/139 (2) — Local
Uveitis (Eye disorders) | 0/136 (0) | 1/139 (1) — Local
Eyelid function disorder (Eye disorders) | 1/136 (1) | 0/139 (0) — Local
Allergic reaction (Immune system disorders) | 0/136 (0) | 1/139 (2) — Local
Other, specify (Surgical and medical procedures) | 4/136 (4) | 2/139 (2) — Local
Other, specify (Ear and labyrinth disorders) | 0/136 (0) | 1/139 (1) — Local
Tinnitus (Ear and labyrinth disorders) | 1/136 (1) | 0/139 (0) — Local
Injection site reaction (General disorders) | 1/136 (1) | 1/139 (1) — Systemic
Fatigue (General disorders) | 70/136 (236) | 69/139 (188) — Systemic
Pain (General disorders) | 3/136 (3) | 4/139 (4) — Systemic
Other, specify (General disorders) | 1/136 (1) | 2/139 (2) — Systemic
Malaise (General disorders) | 30/136 (79) | 28/139 (64) — Systemic
Chills (General disorders) | 29/136 (55) | 29/139 (52) — Systemic
Flu like symptoms (General disorders) | 23/136 (36) | 26/139 (38) — Systemic
Fever (General disorders) | 14/136 (18) | 15/139 (22) — Systemic
Edema limbs (General disorders) | 11/136 (11) | 7/139 (8) — Systemic
Non-cardiac chest pain (General disorders) | 4/136 (4) | 6/139 (7) — Systemic
Irritability (General disorders) | 0/136 (0) | 1/139 (4) — Systemic
Infusion related reaction (General disorders) | 3/136 (3) | 0/139 (0) — Systemic
Localized edema (General disorders) | 0/136 (0) | 1/139 (1) — Systemic
Edema face (General disorders) | 2/136 (2) | 1/139 (1) — Systemic
Edema trunk (General disorders) | 2/136 (2) | 0/139 (0) — Systemic
Gait distrubance (General disorders) | 0/136 (0) | 1/139 (1) — Systemic
Pruritus (Skin and subcutaneous tissue disorders) | 5/136 (5) | 10/139 (12) — Systemic
Other, specify (Skin and subcutaneous tissue disorders) | 14/136 (17) | 10/139 (12) — Systemic
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6/136 (6) | 2/139 (7) — Systemic
Rash acneiform (Skin and subcutaneous tissue disorders) | 6/136 (9) | 4/139 (4) — Systemic
Urticaria (Skin and subcutaneous tissue disorders) | 5/136 (6) | 2/139 (5) — Systemic
Dry skin (Skin and subcutaneous tissue disorders) | 2/136 (2) | 2/139 (3) — Systemic
Nail loss (Skin and subcutaneous tissue disorders) | 1/136 (1) | 2/139 (2) — Systemic
Alopecia (Skin and subcutaneous tissue disorders) | 1/136 (1) | 3/139 (3) — Systemic
Nail ridging (Skin and subcutaneous tissue disorders) | 1/136 (1) | 2/139 (2) — Systemic
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2/136 (2) | 0/139 (0) — Systemic
Nail discoloration (Skin and subcutaneous tissue disorders) | 0/136 (0) | 1/139 (1) — Systemic
Eythema multiforme (Skin and subcutaneous tissue disorders) | 1/136 (1) | 0/139 (0) — Systemic
Arthralgia (Musculoskeletal and connective tissue disorders) | 53/136 (103) | 41/139 (78) — Systemic
Myalgia (Musculoskeletal and connective tissue disorders) | 48/136 (91) | 39/139 (74) — Systemic
Other, specify (Musculoskeletal and connective tissue disorders) | 3/136 (4) | 2/139 (2) — Systemic
Back pain (Musculoskeletal and connective tissue disorders) | 38/136 (85) | 39/139 (58) — Systemic
Bone pain (Musculoskeletal and connective tissue disorders) | 22/136 (47) | 21/139 (47) — Systemic
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12/136 (15) | 13/139 (16) — Systemic
Fracture (Musculoskeletal and connective tissue disorders) | 1/136 (1) | 0/139 (0) — Systemic
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2/136 (2) | 3/139 (5) — Systemic
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 4/139 (4) — Systemic
Neck pain (Musculoskeletal and connective tissue disorders) | 3/136 (3) | 0/139 (0) — Systemic
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2/136 (2) | 0/139 (0) — Systemic
Arthritis (Musculoskeletal and connective tissue disorders) | 1/136 (1) | 1/139 (1) — Systemic
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1/136 (1) | 0/139 (0) — Systemic
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 1/139 (1) — Systemic
Myositis (Musculoskeletal and connective tissue disorders) | 1/136 (1) | 0/139 (0) — Systemic
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1/136 (1) | 0/139 (0) — Systemic
Exostosis (Musculoskeletal and connective tissue disorders) | 0/136 (0) | 1/139 (1) — Systemic
Headache (Nervous system disorders) | 57/136 (158) | 57/139 (146) — Systemic
Other, specify (Nervous system disorders) | 2/136 (2) | 0/139 (0) — Systemic
Dizziness (Nervous system disorders) | 13/136 (15) | 17/139 (25) — Systemic
Neuropathy (Nervous system disorders) | 3/136 (6) | 5/139 (8) — Systemic
Peripheral sensory neuropathy (Nervous system disorders) | 7/136 (8) | 8/139 (8) — Systemic
Dysguesia (Nervous system disorders) | 1/136 (1) | 2/139 (3) — Systemic
Neuralgia (Nervous system disorders) | 3/136 (3) | 2/139 (2) — Systemic
Lethargy (Nervous system disorders) | 0/136 (0) | 2/139 (5) — Systemic
Syncope (Nervous system disorders) | 2/136 (2) | 2/139 (2) — Systemic
Peripheral motor neuropathy (Nervous system disorders) | 1/136 (1) | 1/139 (2) — Systemic
Concentration impairment (Nervous system disorders) | 0/136 (0) | 1/139 (2) — Systemic
Vasovagal reactions (Nervous system disorders) | 0/136 (0) | 1/139 (1) — Systemic
Trigeminal nerve disorder (Nervous system disorders) | 1/136 (1) | 0/139 (0) — Systemic
Somnolence (Nervous system disorders) | 1/136 (1) | 0/139 (0) — Systemic
Seizure (Nervous system disorders) | 0/136 (0) | 1/139 (1) — Systemic
Radiculitis (Nervous system disorders) | 0/136 (0) | 1/139 (1) — Systemic
Presyncope (Nervous system disorders) | 1/136 (1) | 0/139 (0) — Systemic
Paresthesia (Nervous system disorders) | 0/136 (0) | 4/139 (5) — Systemic
Memory impairment (Nervous system disorders) | 0/136 (0) | 1/139 (1) — Systemic
Edema cerebral (Nervous system disorders) | 0/136 (0) | 1/139 (1) — Systemic
Depressed level of consciousness (Nervous system disorders) | 0/136 (0) | 1/139 (1) — Systemic
Nausea (Gastrointestinal disorders) | 38/136 (87) | 38/139 (88) — Systemic
Other, specify (Gastrointestinal disorders) | 8/136 (9) | 3/139 (4) — Systemic
Diarrhea (Gastrointestinal disorders) | 25/136 (48) | 16/139 (29) — Systemic
Abdominal pain (Gastrointestinal disorders) | 8/136 (9) | 7/139 (13) — Systemic
Vomiting (Gastrointestinal disorders) | 9/136 (11) | 10/139 (12) — Systemic
Constipation (Gastrointestinal disorders) | 6/136 (11) | 7/139 (7) — Systemic
GERD (Gastrointestinal disorders) | 4/136 (4) | 7/139 (10) — Systemic
Dyspepsia (Gastrointestinal disorders) | 4/136 (5) | 6/139 (6) — Systemic
Mucositis oral (Gastrointestinal disorders) | 2/136 (2) | 4/139 (5) — Systemic
Bloating (Gastrointestinal disorders) | 2/136 (2) | 2/139 (2) — Systemic
Flatulence (Gastrointestinal disorders) | 1/136 (1) | 2/139 (2) — Systemic
Oral pain (Gastrointestinal disorders) | 1/136 (1) | 1/139 (1) — Systemic
Hemorrhoids (Gastrointestinal disorders) | 0/136 (0) | 2/139 (2) — Systemic
Pancreatitis (Gastrointestinal disorders) | 1/136 (1) | 0/139 (0) — Systemic
Esophageal obstruction (Gastrointestinal disorders) | 0/136 (0) | 1/139 (1) — Systemic
Dry mouth (Gastrointestinal disorders) | 1/136 (1) | 0/139 (0) — Systemic
Colonic hemorrhage (Gastrointestinal disorders) | 1/136 (1) | 0/139 (0) — Systemic
Colitis (Gastrointestinal disorders) | 0/136 (0) | 1/139 (1) — Systemic
Other, specify (Respiratory, thoracic and mediastinal disorders) | 4/136 (4) | 4/139 (4) — Systemic
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 14/136 (19) | 14/139 (19) — Systemic
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15/136 (15) | 18/139 (21) — Systemic
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11/136 (13) | 12/139 (13) — Systemic
Cough (Respiratory, thoracic and mediastinal disorders) | 12/136 (13) | 15/139 (16) — Systemic
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2/136 (2) | 5/139 (8) — Systemic
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5/136 (6) | 4/139 (5) — Systemic
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 3/136 (3) | 0/139 (0) — Systemic
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0/136 (0) | 2/139 (2) — Systemic
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2/136 (2) | 0/139 (0) — Systemic
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0/136 (0) | 1/139 (1) — Systemic
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1/136 (1) | 0/139 (0) — Systemic
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1/136 (1) | 0/139 (0) — Systemic
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 3/136 (3) | 0/139 (0) — Systemic
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1/136 (1) | 0/139 (0) — Systemic
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1/136 (1) | 0/139 (0) — Systemic
Other, specify (Infections and infestations) | 5/136 (6) | 2/139 (2) — Systemic
Upper respiratory infection (Infections and infestations) | 12/136 (16) | 9/139 (12) — Systemic
Sinusitis (Infections and infestations) | 9/136 (12) | 7/139 (10) — Systemic
Urinary tract infection (Infections and infestations) | 6/136 (6) | 5/139 (7) — Systemic
Skin infection (Infections and infestations) | 4/136 (4) | 1/139 (1) — Systemic
Breast infection (Infections and infestations) | 2/136 (2) | 3/139 (3) — Systemic
Skin infection (Infections and infestations) | 3/136 (3) | 2/139 (2) — Systemic
Vaginal infection (Infections and infestations) | 2/136 (3) | 2/139 (2) — Systemic
Lip infection (Infections and infestations) | 2/136 (2) | 1/139 (1) — Systemic
Bronchial infection (Infections and infestations) | 3/136 (4) | 1/139 (1) — Systemic
Otitis media (Infections and infestations) | 2/136 (2) | 1/139 (1) — Systemic
Wound infection (Infections and infestations) | 1/136 (1) | 1/139 (1) — Systemic
Pharyngitis (Infections and infestations) | 1/136 (1) | 0/139 (0) — Systemic
Papulopustular rash (Infections and infestations) | 1/136 (1) | 1/139 (1) — Systemic
Nail infection (Infections and infestations) | 1/136 (1) | 1/139 (1) — Systemic
Mucosal infection (Infections and infestations) | 1/136 (2) | 0/139 (0) — Systemic
Laryngitis (Infections and infestations) | 1/136 (1) | 1/139 (1) — Systemic
Device related infection (Infections and infestations) | 0/136 (0) | 1/139 (1) — Systemic
Bladder infection (Infections and infestations) | 1/136 (1) | 1/139 (1) — Systemic
Tooth infection (Infections and infestations) | 1/136 (1) | 0/139 (0) — Systemic
Paronychia (Infections and infestations) | 0/136 (0) | 1/139 (1) — Systemic
Lung infection (Infections and infestations) | 1/136 (1) | 0/139 (0) — Systemic
Anorectal infection (Infections and infestations) | 0/136 (0) | 1/139 (1) — Systemic
Hot flashes (Vascular disorders) | 16/136 (21) | 18/139 (21) — Systemic
Lymphedema (Vascular disorders) | 9/136 (10) | 7/139 (7) — Systemic
Hypertension (Vascular disorders) | 7/136 (8) | 7/139 (7) — Systemic
Thromboembolic event (Vascular disorders) | 2/136 (2) | 2/139 (2) — Systemic
Hematoma (Vascular disorders) | 2/136 (2) | 0/139 (0) — Systemic
Flushing (Vascular disorders) | 2/136 (2) | 1/139 (1) — Systemic
Superficial thrombophlebitis (Vascular disorders) | 2/136 (2) | 0/139 (0) — Systemic
Peripheral ischemia (Vascular disorders) | 1/136 (1) | 0/139 (0) — Systemic
Hypotension (Vascular disorders) | 1/136 (1) | 0/139 (0) — Systemic
Other, specify (Investigations) | 2/136 (2) | 2/139 (2) — Systemic
White blood cell decreased (Investigations) | 1/136 (2) | 6/139 (8) — Systemic
Ejection fraction decreased (Investigations) | 4/136 (4) | 5/139 (5) — Systemic
Creatinine increased (Investigations) | 1/136 (1) | 4/139 (5) — Systemic
Alanine aminotransferase increased (Investigations) | 2/136 (3) | 3/139 (3) — Systemic
Weight gain (Investigations) | 1/136 (1) | 4/139 (4) — Systemic
Neutrophil count decreased (Investigations) | 0/136 (0) | 4/139 (5) — Systemic
Aspartate aminotransferase increased (Investigations) | 3/136 (3) | 1/139 (1) — Systemic
Lymphocyte count decreased (Investigations) | 0/136 (0) | 3/139 (3) — Systemic
Alkaline phosphatase increased (Investigations) | 1/136 (1) | 2/139 (2) — Systemic
Platelet count decreased (Investigations) | 2/136 (2) | 0/139 (0) — Systemic
Weight loss (Investigations) | 0/136 (0) | 1/139 (1) — Systemic
Chloesterol high (Investigations) | 0/136 (0) | 1/139 (1) — Systemic
Activated partial thromboplastin time prolonged (Investigations) | 0/136 (0) | 1/139 (1) — Systemic
Other, specify (Injury, poisoning and procedural complications) | 2/136 (2) | 1/139 (1) — Systemic
Bruising (Injury, poisoning and procedural complications) | 1/136 (2) | 3/139 (3) — Systemic
Fracture (Injury, poisoning and procedural complications) | 3/136 (3) | 2/139 (2) — Systemic
Fall (Injury, poisoning and procedural complications) | 4/136 (5) | 0/139 (0) — Systemic
Seroma (Injury, poisoning and procedural complications) | 2/136 (2) | 0/139 (0) — Systemic
Spinal fracture (Injury, poisoning and procedural complications) | 1/136 (1) | 1/139 (1) — Systemic
Dermatitis radiation (Injury, poisoning and procedural complications) | 1/136 (1) | 1/139 (1) — Systemic
Burn (Injury, poisoning and procedural complications) | 0/136 (0) | 1/139 (1) — Systemic
Wrist fracture (Injury, poisoning and procedural complications) | 0/136 (0) | 1/139 (1) — Systemic
Wound dehiscence (Injury, poisoning and procedural complications) | 1/136 (1) | 0/139 (0) — Systemic
Radiation recall reaction (Injury, poisoning and procedural complications) | 1/136 (1) | 0/139 (0) — Systemic
Other, specify (Psychiatric disorders) | 1/136 (1) | 1/139 (1) — Systemic
Insomnia (Psychiatric disorders) | 11/136 (13) | 11/139 (11) — Systemic
Anxiety (Psychiatric disorders) | 4/136 (5) | 8/139 (8) — Systemic
Depression (Psychiatric disorders) | 7/136 (7) | 5/139 (5) — Systemic
Agitation (Psychiatric disorders) | 0/136 (0) | 2/139 (2) — Systemic
Personality change (Psychiatric disorders) | 0/136 (0) | 1/139 (1) — Systemic
Libido decreased (Psychiatric disorders) | 1/136 (1) | 0/139 (0) — Systemic
Confusion (Psychiatric disorders) | 0/136 (0) | 1/139 (1) — Systemic
Hyperglycemia (Metabolism and nutrition disorders) | 3/136 (12) | 5/139 (6) — Systemic
Anorexia (Metabolism and nutrition disorders) | 3/136 (3) | 3/139 (3) — Systemic
Hypokalemia (Metabolism and nutrition disorders) | 3/136 (3) | 0/139 (0) — Systemic
Dehydration (Metabolism and nutrition disorders) | 2/136 (3) | 0/139 (0) — Systemic
Hyponatremia (Metabolism and nutrition disorders) | 1/136 (1) | 1/139 (1) — Systemic
Hypocalcemia (Metabolism and nutrition disorders) | 1/136 (1) | 1/139 (1) — Systemic
Hyperkalemia (Metabolism and nutrition disorders) | 0/136 (0) | 2/139 (2) — Systemic
Hypercalcemia (Metabolism and nutrition disorders) | 0/136 (0) | 2/139 (2) — Systemic
Other, specify (Eye disorders) | 4/136 (5) | 1/139 (4) — Systemic
Watering eyes (Eye disorders) | 1/136 (1) | 4/139 (4) — Systemic
Blurred vision (Eye disorders) | 1/136 (6) | 0/139 (0) — Systemic
Floaters (Eye disorders) | 1/136 (1) | 1/139 (1) — Systemic
Conjuctivitis (Eye disorders) | 0/136 (0) | 2/139 (2) — Systemic
Optic nerve disorder (Eye disorders) | 1/136 (1) | 0/139 (0) — Systemic
Dry eye (Eye disorders) | 0/136 (0) | 1/139 (1) — Systemic
Cataract (Eye disorders) | 0/136 (0) | 1/139 (1) — Systemic
Other, specify (Cardiac disorders) | 1/136 (1) | 1/139 (1) — Systemic
Palpitations (Cardiac disorders) | 4/136 (4) | 6/139 (6) — Systemic
Left ventricular systolic dysfunction (Cardiac disorders) | 3/136 (3) | 4/139 (4) — Systemic
Right ventricular dysfunction (Cardiac disorders) | 1/136 (1) | 2/139 (2) — Systemic
Heart failure (Cardiac disorders) | 1/136 (1) | 2/139 (2) — Systemic
Supraventricular tachycardia (Cardiac disorders) | 1/136 (1) | 0/139 (0) — Systemic
Sinus tachycardia (Cardiac disorders) | 0/136 (0) | 2/139 (2) — Systemic
Atrial flutter (Cardiac disorders) | 0/136 (0) | 1/139 (1) — Systemic
Atrial fibrillation (Cardiac disorders) | 0/136 (0) | 1/139 (1) — Systemic
Aortic valve disease (Cardiac disorders) | 1/136 (1) | 0/139 (0) — Systemic
Other, specify (Reproductive system and breast disorders) | 1/136 (3) | 3/139 (3) — Systemic
Breast pain (Reproductive system and breast disorders) | 5/136 (6) | 2/139 (2) — Systemic
Vaginal dryness (Reproductive system and breast disorders) | 5/136 (6) | 1/139 (1) — Systemic
Vaginal hemorrhage (Reproductive system and breast disorders) | 1/136 (3) | 0/139 (0) — Systemic
Vaginal discharge (Reproductive system and breast disorders) | 1/136 (1) | 1/139 (1) — Systemic
Pelvic pain (Reproductive system and breast disorders) | 1/136 (1) | 1/139 (1) — Systemic
Vaginal inflammation (Reproductive system and breast disorders) | 1/136 (1) | 0/139 (0) — Systemic
Dyspareunia (Reproductive system and breast disorders) | 1/136 (1) | 0/139 (0) — Systemic
Urinary tract infection (Renal and urinary disorders) | 1/136 (1) | 3/139 (9) — Systemic
Cystitis noninfective (Renal and urinary disorders) | 2/136 (3) | 1/139 (1) — Systemic
Urinary incontinence (Renal and urinary disorders) | 1/136 (1) | 2/139 (2) — Systemic
Urinary frequency (Renal and urinary disorders) | 1/136 (1) | 2/139 (2) — Systemic
Urinary urgency (Renal and urinary disorders) | 0/136 (0) | 2/139 (2) — Systemic
Hematuria (Renal and urinary disorders) | 2/136 (2) | 0/139 (0) — Systemic
Urinary tract pain (Renal and urinary disorders) | 0/136 (0) | 1/139 (1) — Systemic
Renal calculi (Renal and urinary disorders) | 1/136 (1) | 0/139 (0) — Systemic
Allergic reaction (Immune system disorders) | 7/136 (9) | 6/139 (6) — Systemic
Autoimmune disorder (Immune system disorders) | 0/136 (0) | 1/139 (1) — Systemic
Anaphylaxis (Immune system disorders) | 0/136 (0) | 1/139 (1) — Systemic
Other, specify (Blood and lymphatic system disorders) | 1/136 (1) | 0/139 (0) — Systemic
Anemia (Blood and lymphatic system disorders) | 5/136 (12) | 5/139 (5) — Systemic
Other, specify (Surgical and medical procedures) | 4/136 (5) | 4/139 (4) — Systemic
Tinnitus (Ear and labyrinth disorders) | 2/136 (2) | 1/139 (1) — Systemic
Vertigo (Ear and labyrinth disorders) | 2/136 (2) | 1/139 (1) — Systemic
Hearing impaired (Ear and labyrinth disorders) | 2/136 (2) | 0/139 (0) — Systemic
Ear pain (Ear and labyrinth disorders) | 1/136 (1) | 1/139 (1) — Systemic
Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/136 (1) | 1/139 (2) — Systemic
Other, specify (Endocrine disorders) | 1/136 (1) | 0/139 (0) — Systemic
Hypothyroidism (Endocrine disorders) | 1/136 (1) | 1/139 (1) — Systemic
Hyperthyroidism (Endocrine disorders) | 0/136 (0) | 1/139 (1) — Systemic
Other, specify (Hepatobiliary disorders) | 0/136 (0) | 1/139 (1) — Systemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event a Study is a multi-center clinical study, Institution and Principal Investigator will refrain from any disclosure or publication of Study data until the earlier of: (i) the publication of a multi-center publication or (ii) eighteen months following the conclusion of the Study. Nothing in this Article 6 is intended to limit or restrict in any way Sponsor's right to publish independently any Study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT01570036/Prot_SAP_000.pdf